

## Illuminating nerves, preserving function.™ Precision Surgery.™

3210 Merryfield Row, San Diego, CA 92121

## PHASE 1/2 TRIAL OF ALM-488 IN PATIENTS UNDERGOING HEAD & NECK SURGERY

PROTOCOL NUMBER: ALM-488-001

**Product:** ALM-488 Sterile Solution

**Sponsor:** Alume Biosciences, Inc.

3210 Merryfield Row

San Diego, CA 92121

**Date of Protocol:** 24 August 2020

| Protocol Version | Issue Date |
|-------------------|----------------|
| Original Protocol | 26 April 2020 |
| Amendment 1 | 24 August 2020 |

## **STUDY SUMMARY**

| M-488 Sterile Solution M-488 se 1/2 Trial Of ALM-488 In Patients Undergoing Head & Neck Surgery M-488-001 se 1/2 months lti-center study (United States) mary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. |
|---|
| M-488 se 1/2 Trial Of ALM-488 In Patients Undergoing Head & Neck Surgery M-488-001 se 1/2 months tti-center study (United States) mary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. ondary Objectives: |
| se 1/2 Trial Of ALM-488 In Patients Undergoing Head & Neck Surgery M-488-001 se 1/2 months Iti-center study (United States) nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. |
| se 1/2 Trial Of ALM-488 In Patients Undergoing Head & Neck Surgery M-488-001 se 1/2 months Iti-center study (United States) nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. |
| M-488-001 se 1/2 months tti-center study (United States) nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. ondary Objectives: |
| se 1/2 months tti-center study (United States) mary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. ondary Objectives: |
| nonths Iti-center study (United States) nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. ondary Objectives: |
| ti-center study (United States) nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. Tondary Objectives: |
| nary Objective: To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery. Ondary Objectives: |
| <ul> <li>To evaluate the safety of ALM-488 administered by intravenous (IV) infusion to patients undergoing head and neck surgery.</li> <li>ondary Objectives:</li> </ul> |
| · · |
| <ul> <li>To characterize the pharmacokinetics (PK) of ALM-488 in patients undergoing head and neck surgery.</li> <li>To determine the recommended dose of ALM-488 needed to generate an adequate fluorescence signal in nerves.</li> <li>To evaluate the effect of timing of administration of ALM-488 relative to surgery (e.g., up to 5 hours before surgery) on adequacy of fluorescence nerve labeling.</li> </ul> |
| <ol> <li>study will be conducted in patients who are undergoing head and neck gery. Each subject must meet the following criteria to be enrolled in this by:</li> <li>usion: <ol> <li>The subject has a neoplasm located in the head and neck including parotid neoplasm, thyroid neoplasm, squamous cell carcinoma or an unknown primary with metastases to the cervical lymph node(s) or is undergoing a neck dissection for head and neck neoplasm in an unknown location.</li> <li>The subject's primary surgical treatment is by parotidectomy (superficial or total) or thyroidectomy (unilateral or bilateral) or cervical neck dissection, respectively.</li> </ol> </li> <li>The subject can understand and is willing to sign a written informed consent document.</li> <li>The subject has a life expectancy of at least 6 months.</li> <li>The subject has a total bilirubin within institution's normal laboratory limits.</li> <li>The subject has an aspartate aminotransferase (AST)/serum glutamicoxaloacetic transaminase (SGOT) and alanine aminotransferase (ALT)/serum glutamic-pyruvic transaminase (SGPT) within institution's normal laboratory limits.</li> </ol> |
| 2<br>3<br>2<br>3<br>6 |

- filtration rate (GFR)  $\geq$  60 mL/min/1.73 m<sup>2</sup>.
- 9. The subject, if of childbearing potential, must have a negative urine or serum pregnancy test and be using a medically acceptable form of contraception (e.g., hormonal birth control, intrauterine devices, double-barrier method) or abstinence. The subject, if male, must use a medically acceptable form of contraception (e.g. condom) or abstinence.
- 10. The subject is willing to remain on-site for approximately 23 hours after administration of ALM-488 or, if required, stay overnight after the surgical procedure.
- 11. The subject plans to undergo head and neck surgery.

## Exclusion:

- 1. The subject has had prior radiation or chemotherapy for any prior head and neck neoplasm.
- 2. The subject has had open surgery in the ipsilateral head and neck within 1 year before administration of the investigational product (IP).
- 3. The subject has abnormal cardiac rhythm not controlled with medication, history of stroke within 1 year, history of coronary events within 1 year, and/or heart failure within 1 year before administration of the IP.
- 4. The subject has a history of drug-induced acute tubular necrosis.
- 5. The subject has current evidence of renal disease defined as glomerular filtration rate (GFR) < 60 mL/min/1.73 m<sup>2</sup>.
- 6. The subject has received a systemic investigational drug of any kind for any indication within 6 weeks before administration of the IP.
- 7. The subject is pregnant or breastfeeding.
- 8. The subject has unresolved acute toxicity from prior anti-cancer therapy, as graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0. Alopecia, neuropathy ≤ Grade 2, and other non-acute toxicities are acceptable.
- 9. The subject has a history of fluorescein allergy.
- 10. The subject has a history of severe or steroid dependent asthma.
- 11. Any other criteria deemed by the PI that may prevent the patient from successfully completing the trial.